CLINICAL TRIAL: NCT03997448
Title: Phase II Study of the Combination of Abemaciclib and Pembrolizumab in Locally Advanced Unresectable or Metastatic Gastroesophageal Adenocarcinoma: Big Ten Cancer Research Consortium BTCRC-GI18-149
Brief Title: Abemaciclib and Pembrolizumab in Locally Advanced Unresectable or Metastatic Gastroesophageal Adenocarcinoma: Big Ten Cancer Research Consortium BTCRC-GI18-149
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder decision
Sponsor: Nataliya Uboha (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Nataliya Uboha, Faculty, University of Wisconsin School of Medicine and Public Health, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GI18-149
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Gastroesophageal Cancer; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — pembrolizumab; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abemaciclib and Pembrolizumab (Experimental): Abemaciclib 150mg days 1-21, and Pembrolizumab 200mg IV, Day 1
  Interventions: Drug: Pembrolizumab; Drug: Abemaciclib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg IV
Drug: Abemaciclib — Abemiciclib 150mg PO

SUMMARY:
This study will test the combination of abemaciclib with pembrolizumab in patients with gastric, gastroesophageal junction, or esophageal adenocarcinoma that is metastatic or cannot be surgically removed, and who have progressed on, or were unable to tolerate, at least 2 earlier courses of treatment for their advanced disease.

DETAILED DESCRIPTION:
This is a Phase II non-randomized, single arm, open label study of abemaciclib in combination with pembrolizumab in patients with unresectable or metastatic gastric, gastroesophageal junction, or esophageal adenocarcinoma who have received at least two lines of prior therapy. Treatment will be administered in 21-day cycles. Pembrolizumab will be administered intravenously (IV) at a dose of 200 mg on day 1 of each cycle. Abemaciclib will be taken orally twice a day on each day of the cycle, 150 mg per dose. Treatment will continue until disease progression or development of unacceptable toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic or locally advanced unresectable gastric, gastroesophageal junction or esophageal adenocarcinoma.
* Be willing and able to provide written informed consent for the trial.
* Age >= 18 years at the time of consent.
* Prior treatment with at least two lines of systemic therapy for advanced disease. Patients who have received neoadjuvant or adjuvant therapy or definitive chemoradiation and had recurrence during or within 6 months of completion of all treatments may count adjuvant therapy as one chemotherapy line.
* Presence of measurable disease based on RECIST 1.1 as determined by local site investigator/radiology assessment.
* ECOG PS 0-1.
* Patients must have discontinued all previous treatments for cancer (including cytotoxic chemotherapy, molecularly targeted therapy, radiotherapy, and investigational therapy).
* Patients who received chemotherapy must have recovered (CTCAE Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy. A washout period of at least 21 days is required between last systemic therapy dose and treatment initiation per protocol.
* A washout period of at least 14 days is required between end of radiotherapy and treatment initiation.
* The patient is able to swallow oral medications.
* Demonstrate adequate organ function as defined in the table in the protocol.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 60 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* Men who are not surgically sterile (vasectomy) must agree to use an acceptable method of contraception. Male subjects with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms from the first dose of study drug through at least 60 days after the last dose of study drug. Total abstinence for the same time period is an acceptable alternative.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
* Provided written informed consent and HIPAA authorization for release of personal health information, approved by an Institutional Review Board (IRB). NOTE: HIPAA authorization may be included in the informed consent or obtained separately.

Exclusion Criteria:

* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of prior therapy with CDK4 or CDK6 inhibitors or prior immune checkpoint inhibitors.
* Patients with known microsatellite instability will be excluded.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the study PI.
* Serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Symptomatic central nervous system metastasis. Screening of asymptomatic patients is not required for enrollment.
* Personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Known additional malignancy that progressed or required active treatment within the last 2 years. Exceptions include curatively treated basal cell and squamous cell carcinoma of the skin, curatively resected in situ cervical and/or breast cancers, in situ or intramucosal pharyngeal cancer, and Gleason 6 prostate cancer with PSA <10.
* Patients who have received a live vaccine within 30 days of planned start of pembrolizumab.

Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines, and are not allowed.

* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Active infection requiring systemic therapy.
* Patients who are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 60 days after the last dose of pembrolizumab or abemaciclib. (NOTE: breast milk cannot be stored for future use while the mother is being treated on study.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Uboha, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Univerisy of Iowa Hospital and Clinics, Iowa City, Iowa
  - Rutgers Cancer Institute of NewJjersey, New Brunswick, New Jersey
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Abemaciclib and Pembrolizumab: Pembrolizumab was planned to be administered intravenously (IV) at a dose of 200mg on day 1 of each cycle. Abemaciclib was planned to be administered orally twice a day on each day of the cycle, 150 mg per dose.
Period: Study Treatment
Arm/Group | Abemaciclib and Pembrolizumab
Started | 3
Completed | 1
Not Completed | 2
Not completed — Disease Progression | 1
Not completed — Symptomatic Deterioration | 1
Period: Follow up
Arm/Group | Abemaciclib and Pembrolizumab
Started | 3
Completed | 0
Not Completed | 3
Not completed — Death | 2
Not completed — study terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 68 [46 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status (Baseline) [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 3
    1 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival(PFS)
Description: Progression free survival is defined as the time of treatment initiation until the criteria for disease progression per RECIST1.1 are met or until the date of a death event (any cause). Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From C1D1 until death or up to a maximum of 5 months
Population: Only one subject was assessed per RECIST 1.1 in this trial. Therefore the progression free survival time of only one subject is reported here.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 1
months | NA (NA) — Mean and standard deviation could not be determined due to insufficient number of participants with events.

2. Secondary Outcome: PFS Per irRECIST
Description: A measurement from the date of the start of treatment until the criteria for disease progression is met as defined by irRECIST or death occurs.Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of new lesions is not considered PD but are to be included in the sum diameters. Confirmation required at least 4 weeks after the first irPD assessment provided the patient is considered clinically stable.
Time Frame: From C1D1 until death or up to a maximum of 5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 1
months | NA (NA) — Mean and standard deviation could not be determined due to absence of participants with events.

3. Secondary Outcome: Progression-Free Survival Rate at 6 Months Per RECIST 1.1 and irRECIST
Description: 6 months PFS rate is defined as the proportion of subjects who have experienced no progressive disease or death at a 6 month time point from time of treatment initiation using RECIST and irRECIST criteria. Progressive disease per RECIST 1.1 and irRECIST is defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Per RECIST 1.1, the appearance of one or more new lesions is also considered progression. Per irRECIST, confirmation is required at least 4 weeks after the first irPD assessment provided the patient is considered clinically stable.
Time Frame: From C1D1 until death or up to a maximum of 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 1
months
  RECIST 1.1 | NA (NA) — Mean and standard deviation could not be determined due to insufficient number of participants with events.
  irRECIST | NA (NA) — Mean and standard deviation could not be determined due to absence of participants with events.

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate is the proportion of all subjects with confirmed PR or CR according to RECIST 1.1 and irRECIST criteria, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR/irCR), Disappearance of all target lesions; Partial Response (PR/irPR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From C1D1 until death or up to a maximum of 5 months
Population: Only one subject was assessed per RECIST 1.1 in this trial and only one assessment of PD was recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 1
Participants
  RECIST 1.1 | 0
  irRECIST | 0

5. Secondary Outcome: Disease Control Rate
Description: The disease control rate is the proportion of all subjects with stable disease (SD) for 16 weeks, or partial response (PR), or complete response (CR) according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment). RECIST and irRECIST criteria will be applied. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. Stable disease is defined neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From C1D1 until death or up to a maximum of 5 months
Population: Only one subject was assessed per RECIST 1.1 in this trial and only one assessment of PD was recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 1
Participants
  RECIST 1.1 | 0
  irRECIST | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined by the duration of subject's survival from the start of treatment till death from any cause or off- study.
Time Frame: From C1D1 until death or up to a maximum of 5 months
Measure: Number; unit: months
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 1
months | 1.84

7. Secondary Outcome: Number of Participants With Specified Safety and Tolerability of Abemaciclib in Combination With Pembrolizumab
Description: Safety and tolerability of abemaciclib in combination with pembrolizumab in patients with advanced, unresectable or metastatic gastric, gastroesophageal junction, or esophageal adenocarcinoma, assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: From C1D1 until death or up to a maximum of 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib and Pembrolizumab
Number analyzed (Participants) | 3
Participants
  Number of patients had at least one adverse event of any toxicity grade | 3
  Number of patients had at least one toxicity of grade 3 or greater adverse event | 2
  Number of patients had at least one grade 3 or greater treatment related adverse event | 2
  Number of patients having serious adverse event | 2

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from time of signed informed consent for up to 5 months or until 30 days after discontinuation of study drug(s) or unacceptable toxicity. All-Cause Mortality was assessed from time of signed informed consent for up to 5 months or until death.
Description: An Adverse Event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Abemaciclib and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib and Pembrolizumab (N=3)
DUODENAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
GENERALIZED EDEMA (General disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib and Pembrolizumab (N=3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 2 (3)
ANOREXIA (Metabolism and nutrition disorders) | 2 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
CREATININE INCREASED (Investigations) | 1 (5)
DEPRESSION (Psychiatric disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (2)
EDEMA LIMBS (General disorders) | 1 (1)
FATIGUE (General disorders) | 2 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
THRUSH (Infections and infestations) | 1 (1)
URINE DISCOLORATION (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 1 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT03997448/Prot_SAP_000.pdf